CLINICAL TRIAL: NCT00489515
Title: Visceral Lymphatic Mapping Project: A Pilot Study
Brief Title: Visceral Lymphatic Mapping Using Isosulfan Blue in Patients With Cancer of the Pancreas, Colon, Stomach, Small Intestine, or Gallbladder
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000550095; CCCWFU-99B98; CCCWFU-BG99-047
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-02

CONDITIONS: Colorectal Cancer; Gallbladder Cancer; Gastric Cancer; Pancreatic Cancer; Small Intestine Cancer
Keywords: adenocarcinoma of the gallbladder; stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; stage I gastric cancer; stage II gastric cancer; stage III gastric cancer; stage IV gastric cancer; localized gallbladder cancer; small intestine adenocarcinoma; adenocarcinoma of the colon; adenocarcinoma of the pancreas; adenocarcinoma of the stomach
MeSH Terms: conditions — Colorectal Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with gastrointestinal cancer scheduled for surgery

SUMMARY:
RATIONALE: Diagnostic procedures, such as visceral lymphatic mapping using isosulfan blue, may help find cancer of the pancreas, colon, stomach, small intestine, or gallbladder and find out how far the disease has spread.

PURPOSE: This clinical trial is studying the side effects and how well visceral lymphatic mapping using isosulfan blue works in patients with cancer of the pancreas, colon, stomach, small intestine, or gallbladder.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the safety and feasibility of visceral lymphatic mapping using isosulfan blue in patients with adenocarcinoma of the pancreas, colon, stomach, small bowel, or gallbladder.
* Evaluate the ability of surgically defined sentinel lymph nodes to predict whether other lymph nodes in the basin are involved with the tumor in these patients.

Secondary

* Compare the results obtained from the sentinel lymph node (i.e., positive or negative for metastatic disease) with the results obtained from the other nodes in these patients.
* Compare immunohistochemical analysis with standard analysis of the sentinel lymph nodes in these patients.
* Evaluate the value of intraoperative touch prep analysis of sentinel lymph nodes in these patients.

OUTLINE: This is a pilot study.

During surgical resection of the primary tumor, patients receive isosulfan blue subcutaneously 5 minutes before undergoing sentinel lymph node identification/excision and radical lymphadenectomy. Tissue samples are analyzed by IHC for cytokeratins and CEA.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of adenocarcinoma of 1 of the following sites:

  * Pancreas
  * Stomach
  * Colon
  * Small bowel
  * Gallbladder
* Patients with highly suspicious pancreatic lesions without definitive tissue biopsy are eligible
* No prior uncontrolled visceral malignancy

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No medical comorbidities that would preclude definitive resection
* No known allergies to isosulfan blue

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with gastrointestinal cancer
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 1999-02; Primary Completion 2009-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Safety, as determined by the number of adverse events resulting from procedure | 1 week
  Safety will be assessed by documenting the number of adverse clinical events resulting from the procedure
Ability of surgically defined sentinel lymph nodes to predict whether other lymph nodes are involved with the tumor | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Edward A. Levine, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Result] Hundley JC, Shen P, Shiver SA, Geisinger KR, Levine EA. Lymphatic mapping for gastric adenocarcinoma. Am Surg. 2002 Nov;68(11):931-5. PMID 12455783
- [Result] Levine EA, Shen P, Shiver SA, Waters G, Brant A, Geisenger KR. Intraoperative imprint cytology for evaluation of sentinel lymph nodes from visceral malignancies. J Gastrointest Surg. 2003 Jul-Aug;7(5):687-91. doi: 10.1016/s1091-255x(03)00069-6. PMID 12850683
- [Result] Waters GS, Geisinger KR, Garske DD, Loggie BW, Levine EA. Sentinel lymph node mapping for carcinoma of the colon: a pilot study. Am Surg. 2000 Oct;66(10):943-5; discussion 945-6. PMID 11261621
- [Result] Thomas KA, Lechner J, Shen P, Waters GS, Geisinger KR, Levine EA. Use of sentinel node mapping for cancer of the colon: 'to map or not to map". Am Surg. 2006 Jul;72(7):606-11; discussion 611-2. PMID 16875082